CLINICAL TRIAL: NCT04512612
Title: Can Pan-Colonic Chromoendoscopy (PCC) Improve Adenoma Detection Rate in FIT-Positive-Patients: A Randomized Study
Acronym: PCC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Singapore General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: PCC2019/2831
Record Dates: First submitted 2020-08-10; First posted 2020-08-13 (Actual); Last update posted 2020-08-13 (Actual); Status verified 2020-08

CONDITIONS: Colon Adenoma
Keywords: FIT- positive; Chromoendoscopy; white light endoscopy; adenoma detection rate; advanced adenoma rate; serrated adenoma rate

STUDY DESIGN:
Intervention Model Description: The participants will be randomised to one of the two groups. The first group will undergo colonoscopy evaluation using pan-colonic chromoendoscopy during withdrawal of endoscope. In the second group, colonoscopy evaluation will be performed using high-definition white light endoscopy during withdrawal
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dye based Chromoendoscopy (Active Comparator): The patients enrolled in this group will undergo pan-colonic chromoendoscopy evaluation.
  Interventions: Diagnostic Test: Chromoendoscopy
- High Definition White Light Endoscopy (Active Comparator): The patients enrolled in this group will undergo high definition white light endoscopy based evaluation
  Interventions: Diagnostic Test: High definition white light colonoscopy

INTERVENTIONS:
Diagnostic Test: Chromoendoscopy — Participants randomised to Group A will undergo colonoscopic evaluation using dye-based chromoendoscopy
  Arms: Dye based Chromoendoscopy
Diagnostic Test: High definition white light colonoscopy — Participants randomised to Group B will undergo colonoscopic evaluation using high definition white light endoscopy
  Arms: High Definition White Light Endoscopy

SUMMARY:
Colonoscopy is the technique of choice for evaluation of patients with positive fecal occult blood (FIT). Identification of polyps and their removal has been shown to decrease colorectal cancer incidence rates and mortality. Many endoscopic imaging technologies and devices have been developed to increase adenoma detection (ADR) during screening colonoscopies. They vary in the way they work, and some of the technologies are costly and not widely available. Studies has shown the simple to use pan-colonic chromoendoscopy can improve ADR compared to standard colonoscopy. However, there is little evidence on the utility of pan-colonic chromoendoscopy in asymptomatic individuals undergoing colonoscopy after a positive FIT test. In this randomized study, the investigators aim to compare the utility of chromoendoscopy and high-definition white-light endoscopy in asymptomatic individuals undergoing colonoscopy after a positive FIT test

DETAILED DESCRIPTION:
Eligible subjects with positive screening FIT test referred to the Department of Gastroenterology, Singapore General Hospital will be approached and recruited. The included patients will be randomised to either a) Group A- Chromoendoscopy or b) Group B- high definition white light based evaluation.

Hypothesis:

The investigators hypothesize that application of non-absorbable dye during colonoscopy would enhance the mucosal contrast, delineate the border and surface patterns by accumulating in the innominate grooves and, thereby, enhance the detection of adenoma during colonoscopy

Procedure:

Pan-colonic chromoendoscopy and high-definition white light endoscopy will be performed by five experienced endoscopist, and hospital sedation guidelines will be followed. The colonoscopy will be performed using Olympus (CF-HQ190) or Fujifilm (EC-590) colonoscopies. Indigo carmine dye will be used for pan-colonic chromoendoscopy. Two ampules of Indigo carmine (0.8%, 5ml/ampule) will be dissolved in 250 ml of water and sprayed through the waterjet channel by using the auxiliary foot pump upon reaching the caecum.

The colonoscopy insertion will be performed using high-definition white light, and the scope will be advanced till the caecum. The quality of the bowel preparation will be rated according to the validated Boston bowel preparation score. Participants with inadequate bowel preparation score (Score <6) will be excluded from the study. The fecal residue will be washed, suctioned and cleared during insertion to improve visibility. No special care will be taken to look for lesions during the insertion. Assessment for colonic lesions will only be performed during withdrawal of the endoscope. The minimum withdrawal time was set at 7 minutes. Randomization: Once the caecum is intubated and if the bowel preparation is adequate, the participants will be randomized to pan-colonic chromoendoscopy based withdrawal or high-definition while light based withdrawal. In the pan-colonic chromoendoscopy group, the indigo carmine was sprayed by pressing the auxiliary foot pump, and dye was delivered systematically to coat the entire colonic mucosa. In both, the groups, the lesion size, number, location, morphology will be documented during withdrawal. The investigators characterized the morphology of the lesion according to the established Paris classification. The investigators characterized the lesion as flat neoplasm if the lesion project <2.5mm or polypoid lesion if lesion project >2.5mm into the lumen. The investigators measured the size of the lesions using an open biopsy forceps when needed.

In both the groups, the identified polyps will be removed using the standard techniques, and the tissue will be placed in separate formalin bottles and sent for histology assessment. The histology of the polyps was assessed by dedicated pathologist trained in gastrointestinal pathology. Both the endoscopists and the pathologist will not be blinded to the study technique. The investigators defined advanced adenoma as any adenoma >10 mm in size or with >25% villous histology or high-grade dysplasia. The investigators classified hyperplastic polyps and sessile serrated polyps (SSA) as serrated lesions, The investigators excluded hyperplastic lesions in the rectum from the analysis as such lesions are frequently encountered in the rectum

ELIGIBILITY:
Inclusion Criteria:

* Age older than 50 years
* Positive stool FIT test or FOBT test

Exclusion Criteria:

* Known inflammatory bowel disease
* Known polyposis syndromes
* Previous history of colon cancer and surgical resection
* Overt gastrointestinal bleeding
* Stool FIT or FOBT test performed during hospitalization
* Inadequate bowel preparation (Boston Bowel Preparation score <6 or <2 for each colonic segment)
* Poor patient tolerance to the procedure
* Pregnancy
* Concurrent intake of anticoagulants and thienopyridines (e.g., Clopidogrel), where these drugs cannot be suspended for the adequate duration before colonoscopy
* Patient with known history of hypersensitivity to Indigo carmine dye

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2022-08-01 (Estimated); Study Completion 2022-08-01 (Estimated)

PRIMARY OUTCOMES:
To evaluate the adenoma detection rate between pan-colonic chromoendoscopy and white light colonoscopy | 2 years

SECONDARY OUTCOMES:
Advanced adenoma detection rate white light colonoscopy | 2 years
Flat lesion detection rate | 2 years
Serrated adenoma detection rate | 2 years
Withdrawal time comparison | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Singapore General Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Pohl J, Schneider A, Vogell H, Mayer G, Kaiser G, Ell C. Pancolonic chromoendoscopy with indigo carmine versus standard colonoscopy for detection of neoplastic lesions: a randomised two-centre trial. Gut. 2011 Apr;60(4):485-90. doi: 10.1136/gut.2010.229534. Epub 2010 Dec 15. PMID 21159889
- [Result] Cubiella J, Castells A, Andreu M, Bujanda L, Carballo F, Jover R, Lanas A, Morillas JD, Salas D, Quintero E; COLONPREV study investigators. Correlation between adenoma detection rate in colonoscopy- and fecal immunochemical testing-based colorectal cancer screening programs. United European Gastroenterol J. 2017 Mar;5(2):255-260. doi: 10.1177/2050640616660662. Epub 2016 Jul 20. PMID 28344793